CLINICAL TRIAL: NCT03075098
Title: Diagnostic Accuracy Of Colposcopic Examination in Patients With Oral Dysplastic Lesion (Diagnostic Accuracy Study)
Brief Title: Colposcopy in Detection of Oral Epithelial Dysplasia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sarah badway, assistant lecturer, oral & maxillofacial pathology department, cairo university, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CEBD-CU-2017-03-1
Record Dates: First submitted 2017-03-06; First posted 2017-03-09 (Actual); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Intraepithelial Carcinoma
Keywords: Colposcopy; oral epithelial dysplasia; diagnostic accuracy
MeSH Terms: conditions — Carcinoma in Situ

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- colposcopy of intraepithelial carcinoma (Experimental): Digital colposcope will be used to detect the swede score of the lesion
  Interventions: Device: Digital colposcope

INTERVENTIONS:
Device: Digital colposcope — Diagnostic accuracy of colposcopic examination; Swede scoring system will be used to evaluate the colposcopic examination. Then, the specificity (%) and the sensitivity (%) of colposcopic examination will be calculated using the cutoff value of 8 to segregate dysplastic from non-dysplastic lesions.

SUMMARY:
The aim of this work is to detect the diagnostic accuracy of the intra-oral application of colposcope in diagnosing oral dysplastic lesions in comparison to biopsy taking and histopathological examination.

DETAILED DESCRIPTION:
A- Roles and Responsibilities:

1. The Principle Supervisor: Dr. Mohsen Kazem (M.K.), Professor of Oral &Maxillofacial Pathology, Cairo University, will examine the taken biopsy histopathologically and determine the definitive diagnosis.
2. The Assistant Supervisor: Dr. Heba Dahmoush (H.D.), Professor of Oral & Maxillofacial Pathology, Cairo University, will examine the taken biopsy histopathologically and determine the definitive diagnosis.
3. The Principle Investigator: Sarah Ahmed Mohamed Mahmoud Badawy (S.B.), Assistant Lecturer of Oral &Maxillofacial Pathology, Cairo University, will read and put a colposcopic score for each participant individually.
4. Eman Desouky (E.D.) Sample size calculation; Statistician, Faculty of Oral and Dental Medicine, Cairo University, Egypt.
5. Evidence Based Committee, Faculty of Dentistry, Cairo University: Help in reporting study protocol following STARD guidelines.
6. Ethics Committee, Faculty of Dentistry, Cairo University: Protocol reviewer of the diagnostic accuracy study in order to protect the right, safety, dignity and well-being of the participants.

B- Index test: The principle investigator (S.B.) will perform the index test using Digital Electronic Colposcope (Kernel, KN-2200, China). Before taking up the patients for Colposcopic evaluation and giving them a score, the normal Colposcopic findings will be standardized based on the Colposcopic criteria. Colposcopic criteria includes aceto uptake, surface pattern and clarity of demarcation of the mucosal lesions, vascular pattern, lesion size as well as Iodine staining.

C- Reference test:The reference standard; to reach a definitive diagnosis in oral dysplastic lesions, will be a representative biopsy and histopathological examination. M.K. and H.D. will examine the taken biopsy histopathologically, determine the definitive diagnosis and write the diagnosis in the Assessor chart.

Inclusion criteria:

* Patients seeking for diagnosis of clinically suspected oral dysplastic Leukoplakia or Erythroplakia
* Patients seeking for diagnosis of clinically suspected oral Carcinoma.

Exclusion criteria:

* Patients with secondary infection.
* Patients having other systemic diseases.
* Patients undergoing treatment for the lesions.

ELIGIBILITY:
Inclusion Criteria:

* Patients seeking for diagnosis of clinically suspected oral dysplastic Leukoplakia or Erythroplakia
* Patients seeking for diagnosis of clinically suspected oral Carcinoma.

Exclusion Criteria:

* Patients with secondary infection.
* Patients having other systemic diseases.
* Patients undergoing treatment for the lesions.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2018-01 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of colposcopic examination | Baseline
  using digital colposcope (Kernel, KN-2200, China)

IPD SHARING:
Plan to Share IPD: No